CLINICAL TRIAL: NCT01247402
Title: A Monocenter Randomized Clinical Trial of PAClitaxel drUg-eluting BAlloon Versus Standard Percutaneous Transluminal Angioplasty to Reduce Restenosis in Patients With In-stent Stenoses in the Superficial Femoral and Proximal Popliteal Artery
Brief Title: Paclitaxel Balloon Versus Standard Balloon in In-stent Restenoses of the Superficial Femoral Artery (PACUBA I Trial)
Acronym: PACUBA 1
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Johannes Lammer MD, Professor of Radiology, Department of Radiology, Cardiovascular and Interventional Radiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PACUBA 1
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-10

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; in-stent restenosis; drug eluting balloon
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel eluting balloon (Active Comparator): Freeway 0.035 Paclitaxel eluting balloon (3 microgram Paclitaxel/mm2)
  Interventions: Device: drug eluting balloon angioplasty
- Standard balloon angioplasty (Active Comparator): standard balloon angioplasty
  Interventions: Device: standard balloon angioplasty

INTERVENTIONS:
Device: drug eluting balloon angioplasty — 3 microgram Paclitaxel/mm2 on balloon, 60s application
  Other Names: Freeway 0.035 balloon
  Arms: Paclitaxel eluting balloon
Device: standard balloon angioplasty — standard balloon angioplasty
  Arms: Standard balloon angioplasty

SUMMARY:
Prospective monocenter single-blind randomized (1:1) investigator sponsored clinical trial, in which consecutive patients candidates for percutaneous intervention of angioplasty to treat symptomatic in-stent restenosis of the SFA and P1 segment of the popliteal artery will be assigned to one of two study arms:

1. Treatment Arm: Paclitaxel eluting percutaneous transluminal angioplasty (PePTA)
2. Control Arm: standard percutaneous transluminal angioplasty (sPTA).

Purpose:

To evaluate the morphologic and clinical efficacy of Paclitaxel eluting percutaneous transluminal angioplasty (PePTA) for the reduction of restenosis in SFA and PA stents compared to standard percutaneous transluminal angioplasty (sPTA).

DETAILED DESCRIPTION:
Introduction

Restenosis after endovascular stenting with nitinol stents occurs in up to 30% of the patients at 12 months and up to 50% at 24 months. The rate of recurrence after repeated treatment of SFA in-stent restenoses ranges up to 70% at 6 months.

A recent clinical trial suggested significant inhibition of re-restenosis after treatment of restenosis in coronary stents by Paclitaxel-coated angioplasty balloons.

Study Design

Prospective monocenter single-blind randomized (1:1) investigator sponsored clinical trial, in which consecutive patients candidates for percutaneous intervention of angioplasty to treat symptomatic in-stent restenosis of the SFA and P1 segment of the popliteal artery will be assigned to one of two study arms:

1. Treatment Arm: Paclitaxel eluting percutaneous transluminal angioplasty (PePTA)
2. Control Arm: standard percutaneous transluminal angioplasty (sPTA).

Subject Population:

Consecutive subjects with symptomatic in-stent restenosis of the SFA and P1 segment of the popliteal artery will be screened and enrolled based on the study inclusion and exclusion criteria.

Objectives:

To evaluate the morphologic and clinical efficacy of Paclitaxel eluting percutaneous transluminal angioplasty (PePTA) for the reduction of restenosis in SFA and PA stents compared to standard percutaneous transluminal angioplasty (sPTA).

Primary Endpoints:

Primary patency at 6 month follow up, defined as <50%* diameter stenosis as demonstrated by CDUS and CTA in the absence of clinically driven TLR (Target Lesion Revascularization) during follow-up. Clinically driven TLR defined as reintervention of the target lesion due to presence of a symptomatic >50%* diameter stenosis.

Secondary Endpoints:

1. Technical Success: achievement of a <30%* residual diameter stenosis by visual estimate.
2. Clinical Success: improvement in clinical Rutherford-Becker category after the index procedure.
3. Procedural Success: defined as Device Success without the occurrence of major adverse events (MAE) during the index hospitalization.
4. MAE rate through 30 days post index procedure.
5. Thrombotic occlusion of the Target Lesion at 30 days, 6 months, and 12 months post index procedure.
6. Clinically driven Target Lesion Revascularization (TLR) at 6 months, and 12 months post index procedure.
7. Binary Restenosis rate at 6 month and 12 month FU.

Follow-Up Schedule:

All patients will be followed pre-study, 24 hours post-study, and follow-up evaluations at 30 days, 6 months, and 12 months after the Index procedure. Clinical evaluation and ankle brachial index (ABI) will be assessed pre-study, at 24 hours post-study, and at 6 months, and 12 months after the Index procedure. Colour Doppler ultrasound will be performed at 24 hours post-study, and at 6 months, and 12 months after the Index procedure. Computed tomography angiography (CTA) will be performed at 6 months after the Index procedure.

Study duration:

The enrolment period and follow-up study duration is projected for 24 months.

Subject duration:

Each subject is expected to be enrolled in the study for 12 months.

Inclusion Criteria:

All criteria 1-6 should apply for inclusion.

1. Age > 50 years
2. Patient legally authorized to provide written informed consent
3. Patient willing and likely to comply with the follow up schedule
4. Patient symptomatic Rutherford-Becker 2-5 (Fontaine II-IV)
5. In-stent restenosis in the SFA and P1 segment of the popliteal artery (PA)
6. Tibial run-off of at least 1 artery which however may be stenotic but amenable to PTA

Exclusion Criteria:

1. Patients unable to give informed consent
2. Patients enrolled in another study with any investigational drug or device
3. Major surgical procedures (not including minor amputations) within 30 days prior to this study or planned within 30 days of entry into this study
4. Pregnancy
5. Patients with any known allergy, hypersensitivity or intolerance to radiologic contrast media, ASA, Clopidogrel or Ticlopidine, Paclitaxel
6. Life expectancy of < 1 years

Blood tests:

Total blood count, hematocrit, coagulation parameters, renal function parameters, fibrinogen and hsCRP will be taken before the Index procedure. At 6 months follow up creatinine, fibrinogen and hsCRP will be taken again.

Interventions:

Interventions will be performed percutaneously from an antegrade or an contralateral cross-over approach using 6 French sheaths. Biplane DSA including a ruler fixed at the patients thigh will be performed using two views at least 30° apart to evaluate lesion morphology, inflow disease and run-off. After successful wire passage through the target lesion, patients will be randomly assigned to either Paclitaxel eluting balloon angioplasty (PePTA) or standard percutaneous balloon angioplasty (sPTA) using computer generated random digits and sealed envelopes.

Medical Therapy:

All patients receive aspirin 100mg daily indefinitely and clopidogrel 75 mg daily for 3 months post intervention. Aspirin and clopidogrel will be initiated at least 1 day prior to the intervention, otherwise a loading dose of 300 mg clopidogrel will be given during the intervention.

Control CTA and CDUS:

Angiographic evaluation of restenosis at 6 months will performed using contrast enhanced CTA. At colour Doppler ultrasound evaluation the wave form, peak systolic and diastolic velocity and the peak systolic velocity ration (PSV ratio) will be measured at 24 hours, 6 and 12 months post Index procedure. CDUS findings are consistent with significant restenosis (> 50%), as evidenced by PSV ratio > 2.5 within the treated arterial segment or occlusion of the treated arterial segment.

ELIGIBILITY:
Inclusion Criteria:

All criteria 1-6 should apply for inclusion.

1. Age > 50 years
2. Patient legally authorized to provide written informed consent
3. Patient willing and likely to comply with the follow up schedule
4. Patient symptomatic Rutherford-Becker 2-5 (Fontaine II-IV)
5. In-stent restenosis in the SFA and P1 segment of the popliteal artery (PA)
6. Tibial run-off of at least 1 artery which however may be stenotic but amenable to PTA

Exclusion Criteria:

1. Patients unable to give informed consent
2. Patients enrolled in another study with any investigational drug or device
3. Major surgical procedures (not including minor amputations) within 30 days prior to this study or planned within 30 days of entry into this study
4. Pregnancy
5. Patients with any known allergy, hypersensitivity or intolerance to radiologic contrast media, ASA, Clopidogrel or Ticlopidine, Paclitaxel
6. Life expectancy of < 1 years

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
primary patency rate | 6 months
  Primary patency at 6 month follow up, defined as <50%* diameter stenosis as demonstrated by CDUS and CTA in the absence of clinically driven TLR (Target Lesion Revascularization) during follow-up. Clinically driven TLR defined as reintervention of the target lesion due to presence of a symptomatic >50%* diameter stenosis.

SECONDARY OUTCOMES:
severe adverse events | 30 day

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Lammer, MD, Principal Investigator — Medical Univerity Vienna
Locations (2):
- Austria (2):
  - Angiology, Vienna, Vienna
  - Cardiovascular and Interventional Radiology, AKH-MUW, Vienna, Vienna

REFERENCES:
- [Derived] Kinstner CM, Lammer J, Willfort-Ehringer A, Matzek W, Gschwandtner M, Javor D, Funovics M, Schoder M, Koppensteiner R, Loewe C, Ristl R, Wolf F. Paclitaxel-Eluting Balloon Versus Standard Balloon Angioplasty in In-Stent Restenosis of the Superficial Femoral and Proximal Popliteal Artery: 1-Year Results of the PACUBA Trial. JACC Cardiovasc Interv. 2016 Jul 11;9(13):1386-92. doi: 10.1016/j.jcin.2016.04.012. PMID 27388828